CLINICAL TRIAL: NCT05980689
Title: A Phase II Trial of AK104 Combined With Neoadjuvant Chemoradiotherapy in Proficient Mismatch Repair/Microsatellite Stable Locally Advanced Rectal Cancer
Brief Title: Combination of AK104 and Neoadjuvant Chemoradiotherapy in pMMR/MSS Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Akeso (Industry); Haplox Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, WeiWei Xiao, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2022-766-01
Record Dates: First submitted 2023-07-26; First posted 2023-08-08 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Locally Advanced Rectal Cancer
MeSH Terms: interventions — Capecitabine; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): A total of 33 pMMR/MSS LARC patients will receive long-course chemoradiotherapy plus 2 cycles of AK104, followed by another 3 cycles of AK104, finally received clinical routine manage.
  Interventions: Drug: AK104; Drug: Capecitabine; Radiation: Neoadjuvant Radiotherapy

INTERVENTIONS:
Drug: AK104 — During neo-CRT: 2 cycles of AK104, 10mg/kg d1 q3w. After neo-CRT: 3 cycles of AK104, 10mg/kg d1 q3w.
  Other Names: Cadonilimab
Drug: Capecitabine — During neo-CRT: 825mg/m2 bid Monday-Friday per week
Radiation: Neoadjuvant Radiotherapy — IMRT DT: 50Gy/25Fx

SUMMARY:
This is an open-label, single-arm study to investigate the efficacy and safety of AK104 (an Anti-PD1 and Anti-CTLA4 Bispecific Antibody) and neoadjuvant chemoradiotherapy in patients with pMMR/MSS locally advanced rectal cancer.

DETAILED DESCRIPTION:
The study evaluates the addition of AK104(an Anti-PD1 and Anti-CTLA4 Bispecific Antibody) in neoadjuvant chemoradiotherapy in proficient Mismatch Repair (pMMR) /Microsatellite Stable (MSS) locally advanced rectal cancer (LARC). A total of 33 pMMR/MSS LARC patients will receive long-course chemoradiotherapy plus 2 cycles of AK104, followed by another 3 cycles of AK104, finally received clinical routine manage. The tumor response to treatment, adverse effects and long-term prognosis will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75
2. ECOG 0-1
3. Rectal adenocarcinoma
4. cT3-4aNany or cT1-4aN+
5. No distant metastasis
6. Location ≤12 cm from the anal verge
7. Positive PD-L1 expression (PD-L1 TPS≥1% or PD-L1 CPS ≥1)
8. the MSI status is MSS and pMMR
9. Sufficient bone marrow, kidney and liver function
10. No previous surgery of the rectum, no previous chemotherapy, no previous pelvic radiation, no previous biotherapy, no immunotherapy

Exclusion Criteria:

1. bowel obstruction
2. Distant metastasis
3. Severe arrhythmia, cardiac dysfunction (NYHA grade III or IV )
4. Uncontrollable severe hypertesion
5. Active severe infection
6. Cachexia, organ dysfunction
7. Previous pelvic radiotherapy or chemotherapy
8. Multiple primary cancers
9. Epileptic seizures
10. Malignant history within 5 years, except cervical carcinoma in situ or cutaneous basal cell carcinoma
11. Persons deprived of liberty or under guardianship
12. Impossibility for compliance to follow-up
13. Certain or suspicious allergy to research drug
14. Pregnant or breast-feeding woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | an average of 6 months.
  Rate of complete response (CR), including pathologic complete response (pCR) and clinical complete response (cCR).

SECONDARY OUTCOMES:
Adverse effects | From date of randomization until the date of death from any cause, assessed up to 5 years
  Adverse effects according to CTCAE 5.0
Rate of Major pathologic response and tumor regression grade distribution | an average of 1 year.
  Rate of Major pathologic response and tumor regression grade distribution
Rate of surgical complications | The surgery was scheduled 2-4 weeks after the end of neoadjuvant therapy. And the surgical complications were assessed up to 1 year from the surgery.
  Rate of surgical complications, such as intraoperative hemorrhage, anastomotic leakage, intestinal obstruction, etc.
Disease free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  3 year disease free survival rate
Local recurrence free survival | From date of randomization until the date of first documented pelvic failure, assessed up to 36 months.
  3 year local recurrence free survival rate
Overall survival | From date of randomization until the date of death from any cause, assessed up to 60 months.
  5 year overall survival rate
Long-term anal function | 1.5 year after diagnosis
  Long-term anal function was evaluated using the Wexner Continence Grading Scale ,the score being calculated after the patients' completion of a daily defecatory questionnaire. Range is from 0 (normal continence) to 20 (maximum incontinence with maximum disturbance of lifestyle)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided